CLINICAL TRIAL: NCT06052982
Title: Comparative Randomized Study Evaluating Intra and Postoperative Total Blood Loss During Primary Knee Arthroplasty, With Drainage Versus Non-drainage
Brief Title: Evaluation of Blood Loss During Knee Arthroplasty
Acronym: SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, Dr LHOTELLIER Luc, Orthopedic surgeon, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID RCB : 2019-A01710-57
Record Dates: First submitted 2023-03-23; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Primary Knee Arthroplasty
Keywords: Blood; Loss; Drainage; Without drainage
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (Other): At the end of the knee arthroplasty, a drain is placed at the surgical site
  Interventions: Procedure: Drainage
- Without drain (Other): At the end of the knee arthroplasty, a drain is not placed at the surgical site
  Interventions: Procedure: Drainage

INTERVENTIONS:
Procedure: Drainage — At the end of the knee arthroplasty, a drain is placed or not at the surgical site depending on randomization result

SUMMARY:
Primary arthroplasties are frequent interventions that can present hemorrhagic complications: postoperative hematoma, deglobulization justifying monitoring blood tests and blood transfusion if necessary.

The attitude regarding the drainage of the surgical site supposed to limit these events differs from one surgeon to another, even in the same team. Its use is common practice; for some, systematic. For others, depending on intraoperative findings or the patient's condition. For others, the drain is never laid.

Faced with the divergence of data from the literature on the benefit of the placement of a drain for intra and postoperative bleeding in knee arthroplasty, the lack of randomized prospective studies on large series of patients, and in a desire to homogenization and standardization of the operating procedure of our surgeons, investigators decided to conduct this prospective interventional, comparative and randomized study.

DETAILED DESCRIPTION:
After obtaining the patient's consent and randomisation, the operating surgeon will have the information of placing or not a drain, lately at the end of the intervention so that the course of the intervention is not influenced by the prior knowledge of the patient randomization arm.

Investigators will carry out especially within the framework of this research 3 samples of a total of 10.7 ml of whole blood (appendix. 12.5) distributed as follows:

Sample no. 1 : 2.7 ml of blood in a hemostasis tube (sodium citrate tube) one day before the procedure (D-1) for the determination of the prothrombin level (PT), activated partial thromboplastin time ( TCA) and the INR or International Normalized Ratio.

Sample no. 2 : 4 ml of blood in a purple EDTA tube for NFS, one day before the operation (D-1) for the determination of hemoglobin ( Hb ) and hematocrit ( Hct ) Sample no. 3 : 4 ml of blood in a violet EDTA tube for NFS for the determination of hemoglobin ( Hb ) and hematocrit ( Hct ) on the fifth postoperative day (D5). This last assessment will be prescribed to the patient to be carried out in the rehabilitation center..

The knee prosthesis implantation surgical technique is performed according to the standard operating procedure of the orthopedic surgery team.

According to the operating standard procedure of our orthopedic department, the drain is non-aspirated for 6 hours and then put back under vacuum until the morning after the knee prosthesis operation.

Three months after the intervention the patient will be seen again in consultation and examined.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Patient aged over 18 years
* Patient scheduled for primary knee arthroplasty

Exclusion Criteria:

* Patient expresses his/her opposition to participating in the study
* Patient scheduled for revision, revision or totalization arthroplasty
* Primary arthroplasty after septic arthritis
* Patient requiring an additional planned or unplanned surgical procedure such as TTTA, osteosynthesis for an intraoperative fracture and/or removal of material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin dosage and bleeding quantification in both groups | from the day before surgery until the 5th postoperative day
  Estimation of blood loss with Mercuriali Formula. This formula requires the patient's blood volume and requires the volume of red blood cells transfused as well.

SECONDARY OUTCOMES:
Assessment of blood transfusion during primary knee arthroplasty | from surgery until the 5th postoperative day
  Measurement of total blood transfused between surgery and the fifth day after surgery
Number of patients with complications after knee arthroplasty in the two groups | From surgery up to the third month
  Monitoring for complications from surgery up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Luc LHOTELLIER, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No